CLINICAL TRIAL: NCT02305823
Title: Phase IV Study of the Effectiveness of Aripiprazole, Quetiapine, and Ziprasidone in the Treatment of First Episode of Non-affective Psychosis Individuals Included in the First Episode Psychosis Clinical Program II (PAFIP II)
Brief Title: Comparative Study of Aripiprazole, Quetiapine and Ziprasidone in the Treatment of First Episode Nonaffective Psychosis
Acronym: PAFIP2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Marques de Valdecilla (Other)
Collaborators: Centro de Investigación Biomédica en Red de Salud Mental (Network); Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, Benedicto Crespo-Facorro, Associate Professor of Psychiatry, Fundación Marques de Valdecilla
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZQ2005; CI 2005-0308007 (Other Grant/Funding Number: SENY Fundació Research Grant CI 2005-0308007)
Record Dates: First submitted 2014-11-20; First posted 2014-12-03 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: psychosis; antipsychotic agents; treatment; effectiveness
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Aripiprazole; Quetiapine Fumarate; ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aripiprazole (Active Comparator): Oral, dose range 5-30 mg/day, once or twice a day, during study duration
  Interventions: Drug: Aripiprazole
- Quetiapine (Active Comparator): Oral, dose range 100-600 mg/day, once or twice a day, during study duration
  Interventions: Drug: Quetiapine
- Ziprasidone (Active Comparator): Oral, dose range 40-160 mg/day, once or twice a day, during study duration
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Aripiprazole
  Other Names: Abilify
  Arms: Aripiprazole
Drug: Quetiapine
  Other Names: Seroquel
  Arms: Quetiapine
Drug: Ziprasidone
  Other Names: Zeldox
  Arms: Ziprasidone

SUMMARY:
The selection of antipsychotic in early stages of the illness is mainly determined by its clinical effectiveness. Second generation antipsychotics (SGAs) are the first line drug treatment for individuals suffering from schizophrenia. It is clear that SGAs are not a homogeneous group and clinical effects and profile of side effects differ between SGAs. Differences among antipsychotics in terms of effectiveness have turned out to be a topic of increasing research interest, although comparisons between the different SGAs are scarce. In first episode of psychosis, SGAs have shown a higher treatment effectiveness compared to first generation antipsychotics (FGAs) (findings primarily driven by Haloperidol). Less evident seems to be the notion that some of the SGAs might be more effective (in terms of treatment discontinuation) than others. Most of the medium-term randomized studies have shown similar rates of all-cause treatment discontinuation in first episode patients treated with different SGAs. It may be concluded that more randomized controlled trails should be accomplished to determine the position of frequently used SGAs in clinical practice. The investigators undertook this study with the major objective of comparing the clinical effectiveness of three widely utilized SGAs (Aripiprazole, Ziprasidone and Quetiapine) in the acute treatment of first-episode non-affective psychosis individuals.

DETAILED DESCRIPTION:
Study setting and financial support: data for the present investigation were obtained from an ongoing epidemiological and three-year longitudinal intervention program of first-episode psychosis (PAFIP) conducted at the outpatient clinic and the inpatient unit at the University Hospital Marqués de Valdecilla, Spain. Conforming to international standards for research ethics, this program was approved by the local institutional review board. Patients meeting inclusion criteria and their families provided written informed consent to be included in the PAFIP. The Mental Health Services of Cantabria provided funding for implementing the program. None pharmaceutical company supplied any financial support to it.

Study design: this is a prospective, randomized, flexible-dose, open-label study. At study intake, all patients but eight were antipsychotic naïve. Dose ranges were 5-20 mg /day Aripiprazole, 40-160 mg/day Ziprasidone and 100-600 mg/day Quetiapine. Rapid titration schedule (5-day), until optimal dose was reached, was as a rule used unless severe side effects occur. At the treating physician´s discretion, the dose and type of antipsychotic medication could be changed based on clinical efficacy and the profile of side effects during the follow-up period. Antimuscarinic medication, Lormetazepam and Clonazepam were permitted for clinical reasons. No antimuscarinic agents were administered prophylactically. Antidepressants (Sertraline) and mood stabilizers (lithium) were permitted if clinically needed.

The severity scale of the Clinical Global Impression (CGI) scale, the Brief Psychiatric Rating Scale (BPRS), the Scale for the Assessment of Positive symptoms (SAPS), the Scale for the Assessment of Negative symptoms (SANS), the Calgary Depression Scale for Schizophrenia (CDSS) and the Young Mania Rating Scale (YMRS) were used to evaluate symptomatology. To assess general adverse event experiences the Scale of the Udvalg for Kliniske Undersogelser (UKU), the Simpson-Angus Rating Scale (SARS) and the Barnes Akathisia Scale (BAS) were used. The same trained psychiatrist (BC-F) completed all clinical assessments.

The adverse events were evaluated using the UKU Side effect rating scale. Those treatment-emergent adverse events that occurred at a rate of at least 10% in either treatment group are considered. Treatment-emergent akathisia (BAS) and extrapyramidal symptoms (SARS) were assessed by both baseline-to-end changes and newly emergent categorical changes.

ELIGIBILITY:
Inclusion Criteria:

* 15-60 years.
* Living in the catchment area.
* Experiencing their first episode of psychosis.
* No prior treatment with antipsychotic medication or, if previously treated, a total life time of adequate antipsychotic treatment of less than 6 weeks.
* Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for brief psychotic disorder, schizophreniform disorder, schizophrenia, or schizoaffective disorder.

Exclusion Criteria:

* Meeting DSM-IV criteria for drug dependence
* Meeting DSM-IV criteria for mental retardation
* Having a history of neurological disease or head injury.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 203 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Effectiveness of antipsychotics (percentage of discontinuation of the initially assigned treatment) | 6 weeks
  The main outcomes of effectiveness were the percentage of discontinuation of the initially assigned treatment (patients who completed the 6 weeks follow-up assessment and changed initial antipsychotic) and the mean time to all-cause medication discontinuation. Four reasons for the discontinuation were recorded: 1.- insufficient efficacy; 2.- marked side-effects; 3.- patient reported non-adherence and 4.- other causes. If more than one reason for discontinuation was present, the most important reason according to the above ranking was selected. Data on antipsychotic treatment (doses, discontinuation and concomitant medications) were registered weekly during the first 4 weeks and at 6 week. Insufficient efficacy was established at the treating physician´s judgment only after at least three weeks of treatment.

SECONDARY OUTCOMES:
Change in general psychopathology measured by the Brief Psychiatric Rating Scale (BPRS) | 6 weeks, 3 months and 1 year
  Measured by BPRS. The patients were defined as responders to the optimum dose of antipsychotic at 6 weeks if a >40% reduction of the BPRS scores at intake and had a CGI severity score of ≤ 4. In addition, we also explored to rate of responders if a cutoff of ≥ 50% reduction of the BPRS total scores at intake was used.
Change in positive and negative symptoms measured by the Scale for the Assessment of Negative and Positive Symptoms (SANS and SAPS) | 6 weeks, 3 months and 1 year
  Measured by SANS and SAPS.
Change in the severity of depressive symptoms measured by the Calgary Depression Scale (CDS) | 6 weeks, 3 months and 1 year
  Measured by CDS.
Change in maniac symptoms measured by the Young Mania Rating Scale (YMRS) | 6 weeks, 3 months and 1 year
  Measured by YMRS.
Adherence to treatment | 1 year

OTHER OUTCOMES:
Relapse rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Benedicto Crespo-Facorro, Professor, Principal Investigator — University Hospital Marqués de Valdecilla, IDIVAL, Department of Psychiatry, School of Medicine, University of Cantabria, Santander, Spain. CIBERSAM Centro Investigación Biomédica en Red Salud Mental, Madrid, Spain
Locations (1):
- University Hospital Marques de Valdecilla, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Son J MV, Gomez-Revuelta M, Ayesa-Arriola R, Vazquez-Bourgon J, Foz VO, Ruiz-Veguilla M, Garrido N, Tordesillas-Gutierrez D, Setien-Suero E, Crespo-Facorro B. Comparison of aripiprazole and risperidone effectiveness in first episode non-affective psychosis: Rationale and design of a prospective, randomized, 3-phase, investigator-initiated study (PAFIP-3). Rev Psiquiatr Salud Ment (Engl Ed). 2021 Jul-Sep;14(3):157-163. doi: 10.1016/j.rpsmen.2021.08.002. PMID 34456030
- [Derived] Delgado-Alvarado M, Tordesillas-Gutierrez D, Ayesa-Arriola R, Canal M, de la Foz VO, Labad J, Crespo-Facorro B. Plasma prolactin levels are associated with the severity of illness in drug-naive first-episode psychosis female patients. Arch Womens Ment Health. 2019 Jun;22(3):367-373. doi: 10.1007/s00737-018-0899-x. Epub 2018 Aug 10. PMID 30097769
- [Derived] Tordesillas-Gutierrez D, Ayesa-Arriola R, Delgado-Alvarado M, Robinson JL, Lopez-Morinigo J, Pujol J, Dominguez-Ballesteros ME, David AS, Crespo-Facorro B. The right occipital lobe and poor insight in first-episode psychosis. PLoS One. 2018 Jun 1;13(6):e0197715. doi: 10.1371/journal.pone.0197715. eCollection 2018. PMID 29856773
- [Derived] Pelayo-Teran JM, Gajardo-Galan V, Gomez-Revuelta M, Ortiz-Garcia de la Foz V, Ayesa-Arriola R, Tabares-Seisdedos R, Crespo-Facorro B. Duration of active psychosis and functional outcomes in first-episode non-affective psychosis. Eur Psychiatry. 2018 Aug;52:29-37. doi: 10.1016/j.eurpsy.2018.03.003. Epub 2018 Mar 31. PMID 29614389
- [Derived] Vazquez-Bourgon J, Perez-Iglesias R, Ortiz-Garcia de la Foz V, Suarez Pinilla P, Diaz Martinez A, Crespo-Facorro B. Long-term metabolic effects of aripiprazole, ziprasidone and quetiapine: a pragmatic clinical trial in drug-naive patients with a first-episode of non-affective psychosis. Psychopharmacology (Berl). 2018 Jan;235(1):245-255. doi: 10.1007/s00213-017-4763-x. Epub 2017 Oct 26. PMID 29075885
- [Derived] Ayesa-Arriola R, Alcaraz EG, Hernandez BV, Perez-Iglesias R, Lopez Morinigo JD, Duta R, David AS, Tabares-Seisdedos R, Crespo-Facorro B. Suicidal behaviour in first-episode non-affective psychosis: Specific risk periods and stage-related factors. Eur Neuropsychopharmacol. 2015 Dec;25(12):2278-88. doi: 10.1016/j.euroneuro.2015.09.008. Epub 2015 Sep 28. PMID 26475577